CLINICAL TRIAL: NCT00624013
Title: Effect of Pharmacological Treatment of Depression on A1C and Quality of Life in Underserved Hispanics and African Americans With Diabetes: A Randomized, Placebo Controlled Trial.
Brief Title: Treatment of Diabetes and Depression in Hispanics and African Americans and Its Effect on A1c and Quality of Life.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Charles Drew University of Medicine and Science (Other)
Responsible Party: Principal Investigator, Mayer Davidson, Professor of Medicine, Charles Drew University of Medicine and Science
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 5 U54 RR01616-07
Record Dates: First submitted 2008-02-15; First posted 2008-02-26 (Estimated); Results first posted 2017-12-12 (Actual); Last update posted 2017-12-12 (Actual); Status verified 2017-11

CONDITIONS: Diabetes; Depression
Keywords: Diabetes; Depression; diabetes outcomes; quality of life
MeSH Terms: conditions — Diabetes Mellitus; Depression | interventions — Sertraline

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Placebo (Placebo Comparator): Placebo 50 mg up to 100 mg daily for 6 months
  Interventions: Drug: Placebo
- Sertraline (Zoloft) (Active Comparator): Sertraline (Zoloft) 50 mg up to 100 mg daily for 6 months
  Interventions: Drug: sertraline

INTERVENTIONS:
Drug: sertraline — 50 mg up to 100 mg daily for 6 months
  Other Names: Zoloft
  Arms: Sertraline (Zoloft)
Drug: Placebo — 50 mg up to 100 mg daily for 6 months
  Arms: Placebo

SUMMARY:
This proposed study will test the following hypothesis: Treating depression in Hispanics and African Americans with diabetes will improve their HbA1c and quality of life while on intervention and six months after intervention.

DETAILED DESCRIPTION:
The medication to be used will be sertraline (Zoloft). Sertraline (Zoloft)has been proven in clinical trials to be an effective and well tolerated prescription medication that improves the quality and enjoyment of life for adults suffering from depression . Sertraline is an antidepressant and a member of the family of medications known as selective serotonin reuptake inhibitors (SSRIs). It has excellent tolerability and minimal drug-drug intereactions.

The hypothesis will be tested by the following specific aims:

1. To determine if treating mild to moderate depression with sertraline (Zoloft) in patients with diabetes improves HbA1c.
2. To determine if treating mild to moderate depression with sertraline (Zoloft) in patients with diabetes improves quality of life.

If our hypothesis proves correct and this treatment of depression is efficient and easy in a county hospital population of African Americans and Hispanics, researchers can move forward in finding fast and efficient means of diagnosing depression in vulnerable populations, including low-literate patients. This study is critical in that it stands to improve the HBA1c (and other metabolic parameters) and quality of life of our underserved minority community, which sadly suffers from a higher rate of almost every disease, including diabetes. Treating mild to moderate depression in a county hospital population of African Americans and Hispanics may improve quality of life and reduce/prevent complications and early death. Secondary outcomes include reduced hospitalizations, fewer missed appointments, and improved adherence to medication.

ELIGIBILITY:
Inclusion Criteria:

* All patients (men, women) who are African American or Hispanic over the age of 21 who have been diagnosed with type 2 diabetes and have a HbA1c of greater than 8.0%. Subjects with neuropathic pain will be included in the study. Their pain will be assessed via a validated pain scale. Their primary care providers will treat their pain as necessary.

Exclusion Criteria:

* Pregnant women, patients on dialysis, patients with liver disease or liver enzymes elevated three times above normal, patients with blood pressure greater than 160 systolic or 95 diastolic on two consecutive visits, patients with history of severe depression (as determined by hospitalization or the HAM-D survey) or suicide attempts, patients on therapy for depression, patients already taking SSRI's, and patients with psychotic features or bipolar disease.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 89 (Actual)
Dates: Start 2006-09; Primary Completion 2008-10 (Actual); Study Completion 2008-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mayer Davidson, M.D., Study Director — Charles Drew University School of Medicine
Locations (1):
- Charles Drew University, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Echeverry D, Duran P, Bonds C, Lee M, Davidson MB. Effect of pharmacological treatment of depression on A1C and quality of life in low-income Hispanics and African Americans with diabetes: a randomized, double-blind, placebo-controlled trial. Diabetes Care. 2009 Dec;32(12):2156-60. doi: 10.2337/dc09-0785. Epub 2009 Sep 3. PMID 19729522

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were screened for depression using Whooley's two questions tool at a county diabetes clinic.
Groups:
- Placebo Comparator:Placebo: Placebo: 50 mg up to 100 mg daily for 6 months
- Active Comparator: Sertraline: sertraline: 50 mg up to 100 mg daily for 6 months
Period: Overall Study
Arm/Group | Placebo Comparator:Placebo | Active Comparator: Sertraline
Started | 44 | 45
Completed | 36 | 39
Not Completed | 8 | 6

BASELINE CHARACTERISTICS:
Groups:
- Placebo Comparator: Placebo: Placebo: 50 mg up to 100 mg daily for 6 months
- Total: Total of all reporting groups
Arm/Group | Placebo Comparator: Placebo | Active Comparator: Sertraline | Total
Number analyzed (Participants) | 44 | 45 | 89
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: Eight subjects from placebo arm A dropped the study and six subjects from active comparator group B dropped from the study.
  years
    number analyzed (Participants) | 36 | 39 | 75
    (all) | 53 (10) | 52 (8) | 53 (8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 32 | 33 | 65
  Male | 12 | 12 | 24
Race/Ethnicity, Customized [Number; unit: participants]
  Hispanic | 39 | 39 | 78
  African American | 5 | 5 | 10
Region of Enrollment [Number; unit: participants]
  United States | 44 | 45 | 89

OUTCOME MEASURES:

1. Primary Outcome: HbA1C (%)
Description: Change in HbA1C (%) at month 0 and month 6
Time Frame: Month 0 and month 6
Measure: Mean (Standard Deviation); unit: Percentage of glycosylated hemoglobin
Groups:
- Placebo: Placebo Comparator: 50 mg up to 100 mg daily for 6 months
Arm/Group | Placebo | Sertraline
Number analyzed (Participants) | 36 | 39
Percentage of glycosylated hemoglobin
  HbA1C (%) Month 0 | 9.7 (1.6) | 10.0 (1.8)
  HbA1C (%) Month 6 | 8.8 (1.9) | 8.0 (1.4)

2. Secondary Outcome: Quality of Life
Description: Quality of life (QOL) was assed at baseline and at month 6 using validated instrument Diabetes-39 Quality of Life Questionnaire. It consists of 39-item questionnaire designed to help us learn more about what affects the quality of life of people with diabetes in five dimensions of patients' lives: Diabetes Control, Anxiety and Worry, Social Burden, Sexual Functioning and Energy and Mobility. The Diabetes-39 questionnaire uses a Not Affected At All -Extremely Affected point scale score ranging from 1-7. Raw scale scores were transformed to a 0-100 scale using a linear transformation. Higher values represent a worse outcome. Overall rating of Quality-of-Life was assessed using a Lowest quality-Highest quality scale ranging from 1-7. Higher values represent an increase or improvement in overall QOL. Pattern of Diabetes Severity was measured with a Not Severe at all-Extremely Severe scale ranging from 1-7. Higher values represent increase in diabetes severity.
Time Frame: Month 0 and month 6
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Sertraline (Zoloft)
Number analyzed (Participants) | 36 | 39
units on a scale
  Overall Quality of Life at Month 0 | 3.0 (2) | 3.5 (3)
  Overall Quality of Life at month 6 | 4.0 (2) | 5.0 (3)
  Diabetes Severity at Month 0 | 6.0 (3) | 6.0 (3)
  Diabetes Severity at Month 6 | 5.0 (2) | 5.0 (2)
  Diabetes Control at Month 0 | 66.7 (18.6) | 69.6 (13.4)
  Diabetes Control at Month 6 | 55.7 (17.7) | 49.8 (22.0)
  Anxiety and Worry at Month 0 | 76.7 (16.5) | 78.8 (12.6)
  Anxiety and Worry at Month 6 | 61.9 (22.1) | 57.1 (21.8)
  Social Burden at Month 0 | 63.7 (25.2) | 68.2 (17.3)
  Social Burden at Month 6 | 50.4 (23.8) | 43.8 (25.8)
  Sexual Function at Month 0 | 66.6 (32.4) | 67.8 (28.2)
  Sexual Function at Month 6 | 61.1 (33.2) | 56.7 (31.2)
  Energy and Mobility at Month 0 | 63.1 (20.1) | 67.6 (16.2)
  Energy and Mobility at Month 6 | 49.7 (22.0) | 44.6 (21.1)

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Placebo | Sertraline
Serious Adverse Events (participants affected / at risk) | 2/44 | 0/45
Other Adverse Events (participants affected / at risk) | 1/44 | 3/45
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=44) | Sertraline (N=45)
Suicidal ideation (Psychiatric disorders) | 1 (1) | 0 (0)
skin rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) — subject developed skin rash
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=44) | Sertraline (N=45)
moved out of the country (Social circumstances) | 1 (1) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No